CLINICAL TRIAL: NCT07172087
Title: Construction and Empirical Research of the Applicable Baduanjin Protocol for Patients With Colorectal Cancer Enterostomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Hui Yang, principal investigator, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY-2025-248-02
Record Dates: First submitted 2025-09-02; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Baduanjin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Enterostomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin for patients with enterostomy (Experimental): The validated version of Baduanjin intervention plan for colorectal cancerpatients with enterostomy was adopted, 5 times a week, 15 minutes each time, for 12 weeks.
  Interventions: Other: Baduanjin for patients with enterostomy
- walking exercise (No Intervention): A walking exercise was compared with the version of Baduanjin suitable for enterostomy patients, administered five times a week for 30 minutes each time for 12 weeks.

INTERVENTIONS:
Other: Baduanjin for patients with enterostomy — Modified Baduanjin exercise: a standardized, low-to-moderate intensity qigong regimen consisting of eight sequential movements combined with diaphragmatic breathing. The program excludes any additional resistance or aerobic training and is compared with routine walking exercise only.
  Arms: Baduanjin for patients with enterostomy

SUMMARY:
The goal of this clinical trial is to understand the application effect of the applicable version of Baduanjin protocol in patients with enterostomy and verify the safety and efficacy of this protocol. The main questions it aims to answer are:

Can the applicable version of Baduanjin protocol be safely and effectively applied to patients with enterostomy? Researchers will compare the applicable version of the Baduanjin exercise with the walking exercise to see if the applicable version of the Baduanjin regimen is safe and effective for patients with enterostomy.

Participants will:

Apply the version of Baduanjin exercise or walking exercise five times a week for 12 weeks Patients signed in to the researchers of the project through forms such as exercise record sheets, videos uploaded on wechat, and records made through the keep app.

ELIGIBILITY:
Inclusion Criteria:

1. The disease diagnosis is colorectal cancer
2. At present, enterostomy is used for excretion, and the enterostomy time is more than one month
3. Age ≥ 18 years old
4. Have normal cognitive and expression abilities
5. Voluntarily participate in this study and have signed the informed consent form.

Exclusion Criteria:

1. In the past three months, I have participated in any intervention research or traditional Chinese medical exercise training programs (such as Tai Chi, Baduanjin, other Qigong exercises, etc.)
2. Patients with severe functional disorders of the heart, lungs, liver, kidneys and other organs
3. Mental abnormalities and language expression disorders
4. Patients with limb dysfunction who are unable to cooperate in completing the Baduanjin training
5. Various drainage tubes, PICC catheters, etc. were retained -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Exercise Benefits and Barriers Scale（EBBS） | Baseline (Before enterostomy in patients with colorectal cancer), 4 weeks and 16 weeks after the operation
  This scale consists of two sub-scales with a total of 43 items and two dimensions, namely the benefits of exercise (29 items) and movement disorders (14 items). The Liker 4-level scoring method was adopted, with 1 to 4 points assigned respectively from strongly disagree to strongly agree. The higher the score of the exercise benefit dimension in the calculation dimension, the more exercise benefits the participants perceive. The higher the score of the movement disorder dimension, the more the participants perceive movement disorders.
Pittsburgh Sleep Quality Index（PSQI） | Baseline (Before enterostomy in patients with colorectal cancer) and at 4, 8, 12 and 16 weeks after the operation
  This scale consists of 19 items and 7 dimensions, including subjective sleep quality, time to fall asleep, sleep duration, sleep efficiency, sleep quality, hypnotic drugs, and daytime functional quality, and is used to assess the sleep status of patients in the past month. The Liker 4-level scoring method was adopted, with the maximum total score being 21 points. The higher the score, the poorer the sleep quality of the patient.
Chinese Ostomy Adjustment Inventory（C-OAI） | 4 weeks, 8 weeks, 12 weeks and 16 weeks after enterostomy
  This scale consists of 20 items and 3 dimensions, namely persistent worry (9 items), acceptance (6 items), and a positive attitude towards life (5 items). The scale adopts the Likert 5-point scoring method. Among them, the items with positive implications range from "completely agree" to "completely disagree", with scores ranging from 4 to 0 respectively. Negative meaning items are scored in reverse, ranging from "completely agree" to "completely disagree", with scores ranging from 0 to 4 respectively. The total score of the scale is 80 points. The adaptation level is divided into three grades based on the scale score: < 40 is the low adaptation level, 40-60 is the medium adaptation level, and > 60 is the high adaptation level. The higher the score, the stronger the patient's adaptability to the stoma.
Cancer Fatigue Scale（CFS) | Baseline (Before enterostomy in patients with colorectal cancer) and at 4, 8, 12 and 16 weeks after the operation
  This scale was developed by Okuyama et al. in 2000. It consists of 15 items and is composed of three dimensions: the physical domain (7 items), the emotional domain (4 items), and the cognitive domain (4 items). It uses the Likert 5-level scoring method, ranging from none to very many, with scores ranging from 1 to 5 respectively. The total score ranges from 0 to 60 points. The higher the score, the more severe the patient's fatigue.
Stoma Quality of Life Scale（Stoma-QOL） | 4 weeks, 8 weeks, 12 weeks and 16 weeks after enterostomy
  This scale consists of 20 items, each of which contains 4 options: always, sometimes, rarely, and never, and is assigned a score of 1 to 4 respectively. The patient makes a choice based on their actual situation in the past month. The original score range of the scale is 20 to 80 points, which can be converted to 0 to 100 points. A score of no more than 30 in the quality of life standard is considered the worst level, 31 to 50 is a relatively poor level, 51 to 70 is a relatively high level, and 71 or more is the best level.

OTHER OUTCOMES:
Hemoglobin(Hb) | Baseline (Before enterostomy in patients with colorectal cancer), 5 days after surgery, 4 weeks and 12 weeks after enterostomy
  The protein in red blood cells responsible for transporting oxygen is used to assess anemia or polycythemia; Blood test indicators are collected from the examination results required during the treatment period and do not need to be collected separately outside of the treatment.
Red Blood Cell(RBC) | Baseline (Before enterostomy in patients with colorectal cancer), 5 days after surgery, 4 weeks and 12 weeks after enterostomy
  The most numerous cells in the blood are responsible for carrying oxygen. Abnormal values may indicate anemia, dehydration or bone marrow problems; Blood test indicators are collected from the examination results required during the treatment period and do not need to be collected separately outside of the treatment.
Lymphocyte(LY) | Baseline (Before enterostomy in patients with colorectal cancer), 5 days after surgery, 4 weeks and 12 weeks after enterostomy
  One type of white blood cell, it is an important component of the immune system. An increase or decrease in it may indicate infection, inflammation or immune disease. Blood test indicators are collected from the examination results required during the treatment period and do not need to be collected separately outside of the treatment.
White Blood Cell(WBC) | Baseline (Before enterostomy in patients with colorectal cancer), 5 days after surgery, 4 weeks and 12 weeks after enterostomy
  An increase in the total number usually indicates infection or inflammation, while a decrease may be seen in bone marrow suppression or immune deficiency. Blood test indicators are collected from the examination results required during the treatment period and do not need to be collected separately outside of the treatment.
Prealbumin(PALB) | Baseline (Before enterostomy in patients with colorectal cancer), 5 days after surgery, 4 weeks and 12 weeks after enterostomy
  It is used to assess nutritional status and liver function. A decrease may indicate malnutrition or inflammation. Blood test indicators are collected from the examination results required during the treatment period and do not need to be collected separately outside of the treatment.
Total Protein(TP) | Baseline (Before enterostomy in patients with colorectal cancer), 5 days after surgery, 4 weeks and 12 weeks after enterostomy
  The total sum of all proteins in the plasma, including albumin and globulin, abnormalities may indicate liver disease, kidney disease or immune disorders. Blood test indicators are collected from the examination results required during the treatment period and do not need to be collected separately outside of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Clinical Research Center for Cancer, Sichuan Cancer Hospital & Institute, Sichuan Cancer Center, Afffliated Cancer Hospital of University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No